CLINICAL TRIAL: NCT03508063
Title: Monitoring Physiological Activity Cause by Changes in Physiological Parameters Via Utilization of the Combined Physiological Activity Index (CPAI)
Brief Title: Monitoring Changes in Physiological Parameters by Utilization of the Combined Physiological Activity Index (CPAI)
Status: Completed | Type: Observational
Sponsor: Medasense Biometrics Ltd (Other)
Responsible Party: Sponsor
Other Study IDs: CLI-17-01
Record Dates: First submitted 2018-03-22; First posted 2018-04-25 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy population: Healthy subjects receiving stimuli (thermal stimuli and stressogenic physical stimuli) at rest, and being monitored MCPM.

SUMMARY:
A clinical trial to validate the MCPM (Multi-parameter Combined Physiological Signal-based Monitoring), in estimating physiological activity level, at rest, previous and following stimuli.

DETAILED DESCRIPTION:
The Multi-parameter Combined Physiological Signal-based Monitoring (MCPM) system is a non-invasive multi-parameter physiological monitoring system, intended for continuous . acquisition, analysis and display of physiological signals and a Combined Physiological Activity Index (CPAI).

Subjects who meet the study inclusion and exclusion criteria will be enrolled to the study and their physiological measures, at rest and during exposure to the thermal and stressogenic physical stimuli will be recorded by the MCPM system. All subjects will be recorded according to a standard procedure; subjects will be lying in the supine position and will be instructed to avoid any movements. The experimenter will connect the sensors (MCPM finger probe). During the experimental session, different thermal stimuli will be administrated via the cold pressor test, with 10-20 minutes of non-stimuli interval. The last stimuli is an stressogenic physical preformed by the subject.

1-2 weeks following the first visit, about half of the subjects will be invited to a second visit, identical study visit, to assess the between session test-retest reliability of the signals. During the second visit, CPAI will be measured again under randomize thermal stimuli and an additional 3 Celsius degrees cold stimuli.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 < 65 years old
* Signing an Informed Consent Form (ICF)
* Healthy participant
* No medication/drugs were taken in the last week
* No usage of chronic medication in the last 3 months (except non-pregnancy pills)
* Blood Pressure < (90,140), Heart Rate < 100pps at rest
* No alcohol usage during the last 48 hours

Exclusion Criteria:

* Medication/drugs were taken in the last week (not including non-pregnancy pills)
* Alcohol usage during the last 48 hours
* Caffeine and smoking in the last 3 hours
* Pregnant women
* Inability to comply with the study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy subjects, age: 18-65.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2018-05-21 (Actual)

PRIMARY OUTCOMES:
Performance of the CPAI Index | 6 months
  differentiation between periods in which the subjects were exposed to various intensities of thermal stimuli.

SECONDARY OUTCOMES:
Accuracy of the physiological parameters of the MCPM | 6 months
  comparison to a gold standard device (GE and Procomp system)
Test re-test reliability | 6 months
  comparison of two repeated CPAI and physiological parameters measures of the same individual at two different study visits

CONTACTS AND LOCATIONS:
Overall Officials: Roi Treister, Dr., Principal Investigator — Haifa University, Israel
Locations (1):
- Haifa University, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No